CLINICAL TRIAL: NCT02645643
Title: Intervention to Promote Medical Students Empathy, Well-being and Study emotion-a Randomized Clinical Trial.
Brief Title: Medical Education Intervention for Medical Students
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ming Kuang (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Ming Kuang, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: MEI001
Record Dates: First submitted 2015-12-25; First posted 2016-01-05 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Mental Health
Keywords: medical students; professionalism; medical education; study emotion
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Experimental): Medical students rolled into this group would accept education of medical humanities.
  Interventions: Other: Education of medical humanities
- control group (No Intervention): Medical students rolled into this group would not gain education of medical humanities.

INTERVENTIONS:
Other: Education of medical humanities — The medical students in the intervention group would gain education about the medical humanities, but not the control group.
  Arms: intervention group

SUMMARY:
The doctor-patient relationship was becoming worse. More and more work-related violence has happened to physicians and nurses. A portion of medical students felt depressed and thought that the career future was gloomy. The study was designed to measure the empathy, an vital element of professionalism, well-being of mental and study emotion. Furthermore, the investigators explored an intervention of group study to promote medical students' professionalism, mental health and study emotion.

DETAILED DESCRIPTION:
A total number of 200 junior medical students are going to be enrolled according to inclusive criteria. They are divided into two groups, one group is given education about medical humanities when the other group is not given any intervention but the same room and time.The outcomes including empathy, depression, quality of life, burnout and self-efficiency are measured before, during and after the trial.

ELIGIBILITY:
Inclusion Criteria:

* 1 age 18 to 25 years
* 2 junior students majoring in clinical medicine
* 3 no mental diseases previously

Exclusion Criteria:

* Did not meet inclusion criteria

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Medical students' empathy | 3 months
  we plan to use the scale"The Jefferson Scale of Physician Empathy" to measure medical students' empathy

SECONDARY OUTCOMES:
Medical students' burnout | 3 months
  we plan to use the scale"Maslach Burnout Inventory" to measure medical students' burnout
Quality of life of Medical students | 3 months
  we plan to use the scale"MOS SF-8 Health Survey" to measure medical students' quality of life
Medical students' self-efficiency | 3 months
  we plan to use the "General Self-Efficacy Scale" to measure medical students' self-efficiency
Medical students' depression | 3 months
  we plan to use the "Patient Health Questionnaire-9" to measure medical students' depression

REFERENCES:
- [Background] Schwenk TL, Davis L, Wimsatt LA. Depression, stigma, and suicidal ideation in medical students. JAMA. 2010 Sep 15;304(11):1181-90. doi: 10.1001/jama.2010.1300. PMID 20841531
- [Background] Reed DA, Shanafelt TD, Satele DW, Power DV, Eacker A, Harper W, Moutier C, Durning S, Massie FS Jr, Thomas MR, Sloan JA, Dyrbye LN. Relationship of pass/fail grading and curriculum structure with well-being among preclinical medical students: a multi-institutional study. Acad Med. 2011 Nov;86(11):1367-73. doi: 10.1097/ACM.0b013e3182305d81. PMID 21952063
- [Background] Chen D, Lew R, Hershman W, Orlander J. A cross-sectional measurement of medical student empathy. J Gen Intern Med. 2007 Oct;22(10):1434-8. doi: 10.1007/s11606-007-0298-x. Epub 2007 Jul 26. PMID 17653807
- [Derived] Rong R, Chen W, Dai Z, Gu J, Chen W, Zhou Y, Kuang M, Xiao H. Improvement of the management of mental well-being and empathy in Chinese medical students: a randomized controlled study. BMC Med Educ. 2021 Jul 10;21(1):378. doi: 10.1186/s12909-021-02813-6. PMID 34246265